CLINICAL TRIAL: NCT03094962
Title: Development of Parametric Musculoskeletal Models to Investigate the Anatomy and the Function of the PIP
Brief Title: Development of a Musculoskeletal Model of the PIP Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PUNI1713
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Patient Specific Computational Modeling
Keywords: Kinematics; MRI Scans; CT Scan, Single-Photon Emission; finger interphalangeal joint
MeSH Terms: interventions — Motion Capture; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motion capture, MR scan, CT scan (Other): All volunteers will go through the same data collection process
  Interventions: Other: Motion capture; Diagnostic Test: MR scan; Diagnostic Test: CT scan

INTERVENTIONS:
Other: Motion capture — Capture kinematics of finger movements
Diagnostic Test: MR scan — Capture MR images of hand and fingers in three postures
Diagnostic Test: CT scan — Capture CT images of hand and fingers in three postures

SUMMARY:
The proximal interphalangeal (PIP) joint is the second joint in the finger from the finger tip. The outcome following replacement surgery of this joint is considered unsatisfactory. In order to improve these outcomes, it would be helpful to understand the geometry of the joint, how it moves and the forces that are involved. This can be achieved using computer models that model the bones and the soft tissues - musculoskeletal models. In order to make these models as representative as possible, they should be generated using anatomical data.

Data will initially be extracted from patients' existing magnetic resonance imaging (MRI) and computed tomography (CT) scans. This will enable the computer model to begin being constructed. In parallel to the model initialisation, anatomical and motion data of the PIP joint of healthy volunteers will be collected. The necessary data will be collected using CT and MRI scans, as well as optical motion tracking methods. These data will then be used to populate the musculoskeletal model.

Once the model is constructed, it will be used to simulate the motion of the joint and look at the effect of a simulated PIP joint replacement. This information should then provide insight as to how PIP joint replacements might be improved in future.

ELIGIBILITY:
Inclusion Criteria:

* In general good health
* University of Southampton members of staff
* Over 18 years old and able to provide informed consent
* No known problems relating to the PIP joint

Exclusion Criteria:

* Volunteers involved in other studies concerned with the function and anatomy of the PIP joint which would have adverse effects on this study and/or the study in which they are currently involved.
* Those undergoing treatment related to the PIP joint
* No metallic object should be present in the scanner and therefore those with any implanted metallic devices, or other devices which may cause or be caused adverse effects (e.g. metal plate, pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Capturing hand kinematics using Vicon optical motion capture | 3 years
  Capture hand kinematics of 10 healthy volunteers
Capturing images of the soft tissue in the hand using MR imaging | 3 years
  Capture MR images of the hand for same 10 healthy volunteers as Outcome 1
Capturing images of the bony structures in the hand using CT scanning | 3 years
  Capture CT images of the hand for same 10 healthy volunteers as Outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Christopher WG Phillips, PhD, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams J, Ryall C, Pandyan A, Metcalf C, Stokes M, Bradley S, Warwick DJ. Proximal interphalangeal joint replacement in patients with arthritis of the hand: a meta-analysis. J Bone Joint Surg Br. 2012 Oct;94(10):1305-12. doi: 10.1302/0301-620X.94B10.29035. PMID 23015553